CLINICAL TRIAL: NCT01385007
Title: Preventing Aggression In Veterans With Dementia (PAVED) - Telephone Sub-Study With Rural Veterans
Acronym: PAVED-T
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: South Central VA Mental Illness Research, Education & Clinical Center (U.S. Federal Agency)
Responsible Party: Michael Mallen, PhD, Michael E DeBakey Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-28155
Record Dates: First submitted 2011-06-24; First posted 2011-06-29 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Dementia; Pain
Keywords: Rural; Veterans; Dementia; Pain; Aggression; residence in a VA designated rural area; presence of a caregiver
MeSH Terms: conditions — Dementia; Pain; Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Preventing Aggression in Veterans with Dementia (PAVeD) — PAVeD-Telephone consists of three components: pain-management strategies, improvement of patient-collateral communication skills, and behavioral activation through increased pleasant activity planning. The intervention will be primarily geared toward the caregiver; but patients may be involved in some modules, depending on their dementia severity and willingness. The goal of the sessions is to prevent aggression in veterans with dementia. The sessions will include didactics, skill-building, and discussion. Participants will also be provided a copy of the book, Pain Management for Older Adults: A Self-help Guide, as an additional resource for optional reading on the topics covered in the intervention. The intervention is proposed to include six to eight sessions of weekly treatments, lasting 30 minutes to 45 minutes, specifically developed to address the recognition and management of pain in persons with dementia.

SUMMARY:
Aggression, a common symptom in persons with dementia, is linked with multiple treatable etiologies such as pain, depression, caregiver burden, and caregiver relationships. Pain, the main predictor of aggression, is a common symptom that is inadequately assessed and treated in persons with dementia. The main treatment for aggression is antipsychotic medications that are ineffective, costly, and possess considerable adverse side effects. There is a need to test psychosocial interventions that address treatable causes of aggression. Preliminary data suggest the potential utility of Preventing Aggression in Veterans with Dementia (PAVeD), an evidence-based psychoeducational intervention aimed to prevent aggression, with urban dwelling Veterans. PAVeD, an in-home intervention that requires significant clinician time and expense has yet to be evaluated in a rural culture with Veterans who are in poorer health compared to urban Veterans.

The purpose of this intervention demonstration pilot study is to pilot test and evaluate the PAVeD-Telephone intervention. Twenty rural Veterans with dementia and pain and their caregivers from the Home Based Primary Care (HBPC) Program will be invited to participate. Clinical activities directed toward caregivers are supported by policies and procedures set forth by the Veterans Health Administration (Appendix A). Mixed-methods will be used to collect data using semi-structured interviews and standardized data collection measures suitable for persons with dementia and their caregivers. The interviews go beyond an evaluation of the outcomes by exploring how the intervention was experienced by the dyad.

The specific aims of the study are to:

1. Describe the feasibility and acceptability of the PAVeD-Telephone intervention (number of dyads recruited and completing the study) by rural Veterans and their caregivers.
2. Describe the preliminary outcomes (aggression, depression, Veteran/caregiver relationship quality, pleasant events, caregiver burden, and pain) at baseline, 3 and 6 months.
3. Understand the cultural beliefs and practices of this population and the impact of the intervention.

The PAVeD-Telephone intervention is an innovative approach to shift the paradigm of treating aggression with antipsychotic medications. This study is consistent with the goals of the South Central Mental Illness Research Education and Clinical Center (MIRECC) to improve evidence-based practices in rural Veterans and their caregivers. The next step in this program of research is to submit a Health Services Research and Development Service (HSR&D) application for pilot funding to further develop and test the telephone-based intervention and an appropriate control condition.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of dementia
2. pain symptoms documented by the HBPC staff
3. residence in a VA designated rural area of Lufkin or Conroe
4. presence of a caregiver
5. Enrolled in Home Based Primary Care at Michael E DeBakey VA Medical Center

Exclusion Criteria:

1. display of aggression (spitting, cursing/verbal aggression, hitting, kicking, grabbing, pushing, throwing, biting, scratching, hurting self/others, tearing things/destroying property, making inappropriate verbal sexual advances, or making inappropriate physical sexual advances) in the past year
2. score of 6 or greater on the Functional Assessment Staging (FAST) scale
3. inability to complete by phone a cognitive screening assessment (Telephone Interview for Cognitive Status) or the Philadelphia Geriatric Pain Intensity Scale.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Aggression | 3 months and 6 months post-intervention
  Evaluate the incidence of aggression different than expected in the Telephone PAVeD subjects